CLINICAL TRIAL: NCT01560286
Title: A Phase II, Multi-center, Open-label, Dose-finding Study to Evaluate Safety, Efficacy and Tolerability of Subcutaneously (SC) Administered rAvPAL-PEG in Patients With PKU for 24 Weeks
Brief Title: A Study to Evaluate Subcutaneously Administered rAvPAL-PEG in Patients With Phenylketonuria for 24 Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 165-205
Record Dates: First submitted 2012-03-05; First posted 2012-03-22 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Phenylketonuria
Keywords: PKU; Injections; PEG-PAL; PAL
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): 4-8 week induction of rAvPAL-PEG at 2.5 mg, followed by titration to maintenance dose
  Interventions: Biological: BMN 165 (rAvPAL-PEG)

INTERVENTIONS:
Biological: BMN 165 (rAvPAL-PEG) — Subcutaneous injection of rAvPAL-PEG administered from 1 time up to 5 times per week between 2.5mg up to a maximum of 375mg for 24 weeks.
  Other Names: Recombinant Anabaena variabilis phenylalanine ammonia lyase

SUMMARY:
The primary objective of the study is to evaluate the effect of dosing regimens of multiple subcutaneous (SC) doses of rAvPAL-PEG to induce an early and sustained Phe reduction while decreasing the frequency and severity of hypersensitivity reactions in patients with PKU.

DETAILED DESCRIPTION:
The primary rationale for this study is to define an optimal rAvPAL-PEG dose regimen by establishing the therapeutic effect within the shortest time possible time for induction, titration and maintenance phases while reducing the severity and frequency of hypersensitivity reactions that may lead to dose interruptions. It is hypothesized that these goals can be achieved by keeping rAvPAL-PEG doses low when anti-PEG IgM response is predicted to be high and titrating to an efficacious dose once the IgG response to PAL has developed. Further investigation is needed to determine how early and quickly patients can titrate safely to lower blood Phe; therefore, this protocol proposes to assess two Groups using an induction/titration and maintenance schedule with an aim towards establishing the therapeutic effect safety within an optimal period of time.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of PKU, with the following:

   * Current blood Phe concentration of ≥ 600 µmol/L at Screening.
   * Average blood Phe concentration of ≥ 600 µmol/L over the past 6 months, using available data.
   * Naïve to prior treatment with rAvPAL-PEG.
2. Evidence that the patient is a non responder to Kuvan® treatment (ie, 4 weeks of treatment with 20 mg/kg/day of Kuvan, insufficient response per investigator determination, unsuitable for Kuvan® per Investigator determination, and treatment end date ≥ 2 days prior to Day 1 [ie, first dose]). Patients who have had a previous response to Kuvan® treatment but are not currently taking Kuvan® because of noncompliance and have been off treatment for ≥ 4 months prior to Screening are eligible for participation.
3. Willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures. In the case of participants under the age of 18 or participants who have been deemed mentally unable to provide informed consent, a parent or legal guardian may provide written informed consent (and, if required, the patient will provide written assent).
4. Willing and able to comply with all study procedures.
5. Between the ages of 16 and 70 years, inclusive.
6. Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
7. Sexually active patients must be willing to use an acceptable method of contraception while participating in the study.
8. Maintained a stable diet with no significant modifications during the 4 weeks preceding the administration of study drug and willing to continue with the diet while on study so as to avoid potential variability of response due to variations in dietary intake.
9. In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Exclusion Criteria:

1. Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
2. Use of any medication that is intended to treat PKU, including use of large amino acids, within 2 days prior to the administration of study drug.
3. Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera, within 3 months prior to Screening and during study participation.
4. A prior reaction that included systemic symptoms (eg, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to a PEG containing product. Patients with a prior systemic reaction of generalized rash may be eligible for participation per the discretion of the Principal Investigator in consultation with the Sponsor's Medical Officer.
5. Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.
6. Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
7. Any condition that, in the view of the PI, places the patient at high risk of poor treatment compliance or of not completing the study.
8. Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
9. Creatinine > 1.5 times the upper limit of normal.
10. A positive test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen and hepatitis C antibody.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lounsbury, Study Director — BioMarin Pharmaceutical
Locations (6):
- United States (6):
  - The Children's Hospital, Aurora, Colorado
  - University of Florida, Gainesville, Gainesville, Florida
  - Children's Hospital Boston, Boston, Massachusetts
  - Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - University of Utah Hospital, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BMN 165 (rAvPAL-PEG)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- rAvPAL-PEG: All 24 Enrolled Subjects
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (11.43)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 1
  > or = 18 years | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  Other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Blood Phenylalanine Concentration
Description: All patients will have their plasma Phenylalanine (Phe) assessed. Please note that "Pharmacokinetics Sub-study" was not performed, and thus no results are available.
Time Frame: Baseline, Week 24
Population: The efficacy population will consist of all subjects who received any amount of study drug and have post-treatment blood Phe concentration measurements.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
umol/L
  Baseline | 1168.8 (290.98)
  Week 24 | 617.6 (529.28)

2. Secondary Outcome: Number of Participants With Study Drug Related Adverse Events
Time Frame: Minimum Weekly Assessment of Injection Sites, Vital Signs and Adverse Events. Other Safety Assessments will be performed at other intervals (below):
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Count of Participants; unit: Participants
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
Participants | 23

3. Secondary Outcome: Percentage of Participants With Positive Anti-PAL Immunoglobulin G [IgG]
Description: Antibody Positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 4.3
  Week 24 | 95.5

4. Secondary Outcome: Trough Concentration of BMN 165
Description: PK assessment from pre-dose blood draw.
Time Frame: Week 1, Week 24
Population: The PK population will consist of all subjects who received any amount of study drug and have post-treatment plasma BMN 165 concentration measurements.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
ng/mL
  Week 1 Day 1 | 0.2 (1.09)
  Week 24 | 2341.1 (4768.28)

5. Secondary Outcome: Percentage of Participants With Positive Anti-PEG IgG
Description: Antibody Positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 26.1
  Week 24 | 22.7

6. Secondary Outcome: Percentage of Participants With Positive PAL-IgM
Description: Antibody Positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 34.8
  Week 24 | 90.9

7. Secondary Outcome: Percentage of Participants With Positive Anti-PEG-IgM
Description: Antibody positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 4.3
  Week 24 | 9.1

8. Secondary Outcome: Percentage of Participants With Positive Neutralizing Antibodies [Nab]
Description: Antibody positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 0
  Week 24 | 27.3

9. Secondary Outcome: Percentage of Participants With Positive Anti-PAL-IgE Antibodies
Description: Antibody positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 0
  Week 24 | 0

10. Secondary Outcome: Percentage of Participants With Positive Anti-PAL-PEG IgE Antibodies
Description: Antibody positivity
Time Frame: Baseline, Week 24
Population: The safety population will consist of all subjects who receive any amount of study drug throughout the study duration.
Measure: Number; unit: percentage
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 24
percentage
  Baseline | 0
  Week 24 | 0

ADVERSE EVENTS:
Time Frame: Week 0- Week 24
Arm/Group | rAvPAL-PEG
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAvPAL-PEG (N=24)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAvPAL-PEG (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (9)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Injection site bruising (General disorders) | 10 (13)
Injection site erythema (General disorders) | 13 (40)
Injection site induration (General disorders) | 2 (2)
Injection site pruritus (General disorders) | 5 (11)
Injection site rash (General disorders) | 8 (16)
Injection site reaction (General disorders) | 18 (123)
Injection site swelling (General disorders) | 3 (5)
Injection site urticaria (General disorders) | 2 (3)
Local swelling (General disorders) | 2 (4)
Mass (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 6 (8)
Seasonal allergy (Immune system disorders) | 2 (5)
Nasopharyngitis (Infections and infestations) | 4 (4)
Oral herpes (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 9 (10)
C-reactive protein increased (Investigations) | 3 (3)
Complement factor decreased (Investigations) | 2 (2)
Red blood cell sedimentation rate increased (Investigations) | 2 (2)
Urine albumin/creatinine ratio increased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (80)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (8)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5)
Headache (Nervous system disorders) | 7 (12)
Sinus headache (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 8 (13)
Rash generalised (Skin and subcutaneous tissue disorders) | 5 (10)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (6)
Flushing (Vascular disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days